CLINICAL TRIAL: NCT01311323
Title: Multivessel and Left Main Coronary Artery Stenting in Comparison With Surgical Revascularization in Patients With Non ST Elevation Acute Coronary Syndrome. Prospective, Clinical Randomized Trial (The MILESTONE Trial)
Brief Title: Revascularization Strategies in Patients With Non-ST-Segment Elevation Acute Coronary Syndrome (NSTE-ACS) and Severe Coronary Artery Disease
Acronym: MILESTONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American Heart of Poland (Other)
Collaborators: Andrzej Frycz Modrzewski Krakow University (Other)
Responsible Party: Principal Investigator, Piotr P Buszman, MD, M.D., PhD, Professor, American Heart of Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHP-1
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multivessel Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Multivessel Coronary Artery Disease; Left Main Narrowing; Percutaneous Coronary Intervention; Coronary Artery Bypass Grafting; Drug-Eluting Stent; Fractional Flow Reserve; Instant wave-free ratio; virtual Fractional Flow Reserve
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI with DES implantation (Experimental): Percutaneous Coronary Intervention Implantation of Drug-Eluting Stents
  Interventions: Procedure: PCI
- CABG (Active Comparator): Coronary Artery Bypass Grafting.On-pump or Off-pump CABG
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: PCI — Percutaneous Coronary Intervention with contemporary drug eluting stent, fractional flow reserve or iFR measurement and optimisation with intravascular imaging
  Other Names: •Percutaneous coronary intervention; •Multivessel coronary disease; •Left main narrowing
  Arms: PCI with DES implantation
Procedure: CABG — Coronary Artery Bypass Graft
  Other Names: Multivessel coronary artery disease; Coronary artery bypass graft; Left Main narrowing
  Arms: CABG

SUMMARY:
MILESTONE STUDY is dedicated to problems connected with patients with multivessel coronary artery disease and/or with left main narrowing who present symptoms of acute ischemia. For such kind of patients according to current ACC/AHA guidelines CABG (surgical revascularization) is recommended as a treatment method. In comparison with CABG, recent studies have shown that PCI (percutaneous coronary intervention) is associated with a lower rate of periprocedural adverse events and similar long term event-free survival in patients with left main disease. Our latest non randomized registry and randomized LEMANS study, comparing LMCA (left main coronary artery) stenting with CABG confirmed above findings. LEMANS ACS (acute coronary syndrome) retrospective registry of patients with UPLMCA (unprotected LMCA) disease and non ST elevation ACS showed lower 30 day and trend toward lower one year mortality after PCI when compared with CABG. It should be stressed, that acute ischemia substantially increase the risk of CABG. In fact, there are limited data on the outcome of ULMCA stenting or CABG in patients with acute coronary syndromes (ACS).

Similarly, all randomized studies comparing PCI vs CABG in multivessel disease included mainly patients with stable angina, small cohort of patients with unstable angina and they excluded patients with non ST elevation Myocardial infarction.

In the SYNTAX study -largest PCI vs CABG trial, randomized patients were patients with low perioperative risk (logistic EUROSCORE <5) and ACS patients routinely excluded. High perioperative risk patients were included only in PCI registry.

DETAILED DESCRIPTION:
Within last decade, aging of the population and coexistence of multiple comorbidities influenced a risk of patients presenting with acute coronary syndrome (ACS). Furthermore, a steady decline in ST elevation ACS incidence and increase in non-ST elevation acute coronary syndrome (NSTE-ACS) has been observed, associated with poorer long term prognosis. This is related to the complexity of coronary artery disease in patients with NSTE-ACS, as nearly half of them have multivessel disease (MVD). The optimal revascularization strategy in this group of patients remains unknown. Due to clinical presentation in most of cases early or delayed invasive strategy is preferred by both American and European guidelines, however the method of revascularization is not specified. Due to high surgical risk presentation, immediate stenting of the culprit lesion and delayed complete percutaneous revascularization is becoming a common practice. On the other hand, basing on the anatomical criteria coronary artery bypass grafting (CABG) should be the standard of care . Very few reports addressed so far the problem of optimal revascularization strategy in patients presenting with MVD and NSTE-ACS. A hypothesis of a positive outcome can be derived from some previous studies comparing PCI and CABG in which most of patients enrolled presented with NSTE-ACS, including our experience.

Aim and hypothesis:

Hence, the purpose of this study will be to compare contemporary coronary angioplasty with coronary artery bypass grafting in a prospective, clinical, multicenter, randomized trial. The hypothesis of this study is the non-inferiority of PCI compared to CABG in terms of the primary composite endpoint (death, myocardial infarction, stroke).

Method:

Patients with multivessel coronary artery disease, left main and acute coronary syndrome without ST segment elevation, qualified for early invasive treatment, with a Syntax Score below 33, and in whom the invasive cardiologist and cardiac surgeon will recognize both PCI and CABG as possible to achieve complete revascularization will be enrolled to the study. In the case of centers without the Cardiac Surgery Department, "Heart Team" consultations will take place via videoconference, and records of coronarography and echocardiography will be shared via the PACS (ang. Picture Archiving and Communication System system). The main exclusion criteria will be the qualification for conservative treatment, surgery other than CABG due to structural heart defect, ST segment elevation myocardial infarction, stable coronary artery disease, immediate need for PCI. After fulfilling the inclusion criteria and lack of exclusion criteria, the patient will be randomized in a 1: 1 ratio to either PCI or CABG. The PCI procedure will be performed after assessing the hemodynamic significance of all lesions with vFFR, FFR or iFR or using the latest generation drug eluting stents, and the implantation will be optimized based on intravascular imaging. CABG procedures will be performed based on the experience of the respective center, including the OPCAB technique, and the internal mammary artery will be used in each case. The primary endpoint of the study will be all cause death, myocardial infarction, and stroke in one-year follow-up. To prove the assumed hypothesis of the study, with the test power of 80% alpha error 5% and the percentage of lost to follow-up at the level of 5%, the study should include 500 patients in each group. Secondary endpoints will be ischemia driven revascularization, left ventricular ejection fraction, major and minor bleeding incidence, new onset of atrial fibrillation, de novo heart failure, unscheduled re-hospitalization, quality of life, and cost effectiveness. After the hospitalization, patients will be subjected to strict secondary prevention principles, including cardiac and cardiac surgery rehabilitation, and will undergo four specialistic follow-up visits with cardiac echo and stress tests at selected time points.

Anticipated outcomes:

In the case of positive results of the study, the efficacy and safety of PCI in the studied group of patients will be confirmed. This will contribute to the creation of a new guidelines in a given area, translating into faster and easier access to rapid invasive treatment. It will also facilitate the decision-making process in centers without cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the inclusion criteria to be considered for the trial. If ANY of the exclusion criteria are met, the subject is excluded from the trial and cannot be randomized.

* Age over 18 years,
* Written patient consent,
* Acute Coronary Syndrome without ST-segment elevation of very high, high, and intermediate risk including NSTEMI and unstable angina requiring urgent (within 72 hours) invasive strategy,
* Qualification for invasive treatment,
* Multivessel coronary disease, defined as angiographic narrowing >50%DS in at least two arteries, including involvement of the proximal segment of the left anterior descending artery or three-vessel disease with a Syntax Score < 33. For borderline stenoses (40-70%), vFFR, FFR, or iFR will be decisive,
* Left main coronary artery disease defined as narrowing >50%DS. For borderline changes, IVUS (MLA <6 mm2 or vFFR, FFR, or iFR) with a Syntax Score < 32 will be decisive,
* Feasibility of complete revascularization on both the CABG and PCI sides,
* Consent within the Heart Team for both CABG by the cardiothoracic surgeon and PCI by the interventional cardiologist.

Exclusion Criteria:

* Age under 18 years,
* ST-segment elevation myocardial infarction (STEMI) or new left bundle branch block (LBBB),
* Stable coronary syndrome,
* Single- or two-vessel coronary disease without involvement of the proximal LAD, defined as narrowing above 50%DS,
* Qualification for conservative treatment,
* Anticipated surgery other than CABG due to severe valvular defect or other structural defect, particularly moderate or severe mitral regurgitation,
* Need for immediate coronary angioplasty treatment,
* Syntax Score above 33,
* Contraindications to short-term and long-term antiplatelet therapy,
* Acute heart failure in class IV (cardiogenic shock),
* Previous CABG procedure,
* Previous PCI procedure within the last 6 months,
* Ischemic or hemorrhagic stroke within 6 months prior to inclusion,
* End-stage chronic kidney disease on dialysis,
* Pregnancy or intention to become pregnant (women of child bearing age must have a recent negative pregnancy test prior to randomization),
* Non cardiac co-morbidities with life expectancy less than 3 years,
* Participation in other clinical trial that have not reached their primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
MACCE - Major Adverse Cardiac and Cerebral Events | One year after revascularization procedure
  The primary endpoint is a composite of all cause death, revascularization procedure: PCI or CABG. The hypothesis test is designed to show non-inferiority of PCI to CABG for the primary endpoint

SECONDARY OUTCOMES:
SAE - Serious Adverse Events | peri-hospital period, one month and one year and two years after revascularization procedure
  ischemia driven revascularization, left ventricular ejection fraction, major and minor bleeding incidence, new onset of atrial fibrillation, de novo heart failure, unscheduled re-hospitalization
Procedural and post procedural complication | peri-hospital period, one month and one year after revascularization procedure
  Procedural and post procedural complication: length of hospital stay and frequency of prolonged hospitalization ; return to work; readmissions and cause of readmissions; angina and functional status; medications.
Overall costs of treatment strategies. | one year ofter revascularization procedure
  Hospital costs and long-term cost-effectiveness.
Occurence of stent thrombosis or graft occlusion | peri-hospital period, one month and one year after revascularization procedure
  Stent trombosis will be defined in accordance with ARC definition.
Hemorrhagic complications. | peri-hospital period, one month and one year after revascularization procedure
  Hemorrhagic complications will be clasified according to TIMI scale.
Frequency and impact of complete revascularization | one year after revascularization procedure
  Complete revascularization will be defined on an anatomic basis and by revascularization of all significant ischemic areas.
LVEF | 6 and 12 months
  Left Ventricle Ejection Fraction

CONTACTS AND LOCATIONS:
Overall Officials: Piotr P Buszman, MD,PhD, Prof, Principal Investigator — American Heart of Poland; Krzysztof Sanetra, MD, PhD, Principal Investigator — American Heart of Poland
Locations (5):
- Poland (5):
  - Małopolska Cardiovascular Center, Polish-American Heart Clinic in Chrzanów, Chrzanów, Malopolska
  - Polish-American Heart Clinics Center for Cardiology and Cardiac Surgery Outpatient Specialist Care in Bielsko-Biała, Bielsko-Biala, Silesian Voivodeship
  - Polish-American Heart Clinics III Department of Invasive Cardiology, Angiology and Electrocardiology, Dąbrowa Górnicza, Silesian Voivodeship
  - Polish-American Heart Clinics, 1st Department of Cardiology and Angiology in Ustroń, Ustroń, Silesian Voivodeship
  - Polish-American Heart Clinics X Department of Invasive Cardiology, Electrophysiology and Electrostimulation in Tychy, Tychy

REFERENCES:
- [Background] Park DW, Kim YH, Yun SC, Lee JY, Kim WJ, Kang SJ, Lee SW, Lee CW, Kim JJ, Choo SJ, Chung CH, Lee JW, Park SW, Park SJ. Long-term outcomes after stenting versus coronary artery bypass grafting for unprotected left main coronary artery disease: 10-year results of bare-metal stents and 5-year results of drug-eluting stents from the ASAN-MAIN (ASAN Medical Center-Left MAIN Revascularization) Registry. J Am Coll Cardiol. 2010 Oct 19;56(17):1366-75. doi: 10.1016/j.jacc.2010.03.097. PMID 20946993
- [Background] Park DW, Seung KB, Kim YH, Lee JY, Kim WJ, Kang SJ, Lee SW, Lee CW, Park SW, Yun SC, Gwon HC, Jeong MH, Jang YS, Kim HS, Kim PJ, Seong IW, Park HS, Ahn T, Chae IH, Tahk SJ, Chung WS, Park SJ. Long-term safety and efficacy of stenting versus coronary artery bypass grafting for unprotected left main coronary artery disease: 5-year results from the MAIN-COMPARE (Revascularization for Unprotected Left Main Coronary Artery Stenosis: Comparison of Percutaneous Coronary Angioplasty Versus Surgical Revascularization) registry. J Am Coll Cardiol. 2010 Jul 6;56(2):117-24. doi: 10.1016/j.jacc.2010.04.004. Epub 2010 May 6. PMID 20451344
- [Background] Buszman PE, Buszman PP, Kiesz RS, Bochenek A, Trela B, Konkolewska M, Wallace-Bradley D, Wilczynski M, Banasiewicz-Szkrobka I, Peszek-Przybyla E, Krol M, Kondys M, Milewski K, Wiernek S, Debinski M, Zurakowski A, Martin JL, Tendera M. Early and long-term results of unprotected left main coronary artery stenting: the LE MANS (Left Main Coronary Artery Stenting) registry. J Am Coll Cardiol. 2009 Oct 13;54(16):1500-11. doi: 10.1016/j.jacc.2009.07.007. Epub 2009 Aug 21. PMID 19699048
- [Background] Buszman PP, Bochenek A, Konkolewska M, Trela B, Kiesz RS, Wilczynski M, Cisowski M, Krejca M, Banasiewicz-Szkrobka I, Krol M, Kondys M, Wiernek S, Orlik B, Martin JL, Tendera M, Buszman PE. Early and long-term outcomes after surgical and percutaneous myocardial revascularization in patients with non-ST-elevation acute coronary syndromes and unprotected left main disease. J Invasive Cardiol. 2009 Nov;21(11):564-9. PMID 19901409
- [Background] Buszman PE, Kiesz SR, Bochenek A, Peszek-Przybyla E, Szkrobka I, Debinski M, Bialkowska B, Dudek D, Gruszka A, Zurakowski A, Milewski K, Wilczynski M, Rzeszutko L, Buszman P, Szymszal J, Martin JL, Tendera M. Acute and late outcomes of unprotected left main stenting in comparison with surgical revascularization. J Am Coll Cardiol. 2008 Feb 5;51(5):538-45. doi: 10.1016/j.jacc.2007.09.054. PMID 18237682